CLINICAL TRIAL: NCT00656916
Title: Randomized Study of Early Treatment With Inhaled Corticosteroids Versus Observation for Patients Who Have Decreased Lung Function Status Post Allogeneic Stem Cell Transplantation
Brief Title: Inhaled Corticosteroids Versus Observation for Patients With Decreased Lung Function Status
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0390
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Bronchiolitis
Keywords: Post-Transplant Constrictive Bronchiolitis; Bronchiolitis; Fluticasone Propionate; Inhaled Corticosteroids; Lung Condition; PTCB
MeSH Terms: conditions — Bronchiolitis | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Propionate (Experimental): 440 micrograms twice daily by oral inhalation.
  Interventions: Drug: Fluticasone Propionate
- Observational Group (No Intervention): Comparator group, no intervention.

INTERVENTIONS:
Drug: Fluticasone Propionate — 440 micrograms twice daily by oral inhalation.
  Arms: Fluticasone Propionate

SUMMARY:
The goal of this clinical research study is to compare lung function of patients who inhale steroids in the early stages of post-transplant constrictive bronchiolitis (PTCB) to patients who continue with standard of care.

DETAILED DESCRIPTION:
The Study Drug:

Fluticasone propionate is designed to stop the inflammatory action of asthma cells in PTCB.

Screening Tests:

Before you can start treatment on this study, you will have a pulmonary function test (PFT). For this tests, you will be asked to breathe in several different ways while you have a mouthpiece in your mouth to test your lung function.

Study Groups:

If you are found eligible to take part in this study, participants will be assigned to receive fluticasone propionate.

Study Drug Administration:

You will receive fluticasone propionate twice a day by oral inhalation. The study drug will be taken through a metered-dose inhaler. You will be given detailed instructions by the research nurse or clinic nurse at your first study visit.

You will use an Albuterol MDI (rescue inhaler) when needed for shortness of breath. This inhaler is commonly used to treat asthma, chronic obstructive pulmonary disease (COPD), and other respiratory problems. Your clinic nurse will tell you how to use it.

You will fill out a diary to record how often you use the rescue inhaler. You will also record when you take the study drug each week. The diary will be collected at each visit. The diary will take a few minutes to fill out.

Study Visits:

On Day 1, the following tests and procedures will be performed:

* You will have a 6-minute walk test. To perform the 6-minute walk test, you will walk as far as possible around cones on a flat indoor course that is about 40 yards long. You will walk at your own pace and can take breaks at any time. After 6 minutes, the study staff will check the total distance you have walked. Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be measured before and after the walk. Your oxygen saturation levels will be checked throughout the test. To measure oxygen saturation, you will wear a small clip on your finger that will send the oxygen saturation data to a small computer.
* You will also complete St. George's respiratory questionnaire.The questionnaire will have 17 multiple choice or true/false questions about your lung function and overall health. A research nurse will be available to help you with the questionnaire. It will take about 30 minutes to complete.
* You will also complete a NIOX flex test. This measures the amount of nitric oxide in your lungs. While seated, you will exhale and then place the NIOX filter in your mouth. You will then inhale to full lung capacity over 2-3 seconds. Then you will exhale slowly keeping constant flow with the aid of a meter on the computer screen. This is repeated until 3 valid readings are measured and then the test is completed.

Between Weeks 4 and 6, you will have a PFT.

At 3 months, 6 months, and 1 year, the following tests and procedures will be performed:

* You will have a PFT.
* You will complete the St. George's respiratory questionnaire.
* You will have a 6-minute walk test.
* You will have an exhaled nitric oxide (NIOX) Flex test, only at baseline, 3 and 6 months.

Length of Study:

You will be taken off study if the disease gets worse or if intolerable side effects occur. All patients whose condition stayed the same or improved at the end of 1 year will continue study drug and visit schedule.

End-of-Study Visit:

Before you are considered off-study, you will have an end-of-study visit. The following tests and procedures will be performed:

* You will have a PFT.
* You will complete the St. George's respiratory questionnaire.
* You will have a 6-minute walk test.

Follow-Up:

Patients may be contacted by mail or by phone to answer follow-up questions. Follow-up questions and contact frequency will be based on your condition. If you are contacted by phone, the conversation will last about 15 minutes.

This is an investigational study. Fluticasone propionate is FDA approved and commercially available for use in asthma and COPD patients. It's use in PTCB is investigational. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >/=18 years of age.
2. Patients must be engrafted and at least 80 days post allogeneic hematopoietic stem cell transplantation.
3. New onset airflow obstruction defined as decline of forced expiratory volume in 1 second (FEV1) percent predicted >/= 15%.
4. Total Lung Capacity (TLC) > 85% to rule out restrictive lung disease.
5. Patient must be willing to comply with all study procedures and capable of signing informed consent.

Exclusion Criteria:

1. Patients with active pulmonary infection.
2. Patients with known hypersensitivity to corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Bashoura, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 03/24/08 through 12/15/10. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated due to slow accrual.
Groups:
- Observation: Comparator group, no intervention.
Period: Overall Study
Arm/Group | Fluticasone Propionate | Observation
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate | Observation | Total
Number analyzed (Participants) | 1 | 0 | 1
Age Continuous [Median (Full Range); unit: years] | 46 (0) [46 to 46] |  | 46 [46 to 46]
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Lung Function Non-deterioration Rate
Description: Lung function non deterioration rate defined by change of forced expiratory volume in one second (FEV1) of < 20%. FEV1, maximal amount of air forcefully exhaled in 1 second, converted to percentage of normal, calculated from a pulmonary function test (PFT) performed at baseline and three months.
Time Frame: Baseline and three months
Population: There was no analysis performed for the protocol due the low enrollment (one participant).
Measure: Number; unit: Percentage (FEV1
Arm/Group | Fluticasone Propionate | Observation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fluticasone Propionate | Observation
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes